CLINICAL TRIAL: NCT03555578
Title: Specified Drug-Use Survey of Leuprorelin Acetate Injection Kit 11.25 mg "All-Case Investigation: Spinal and Bulbar Muscular Atrophy (SBMA)"
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Leuprorelin-5004; JapicCTI-183981 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Spinal and Bulbar Muscular Atrophy
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked | interventions — Leuprolide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Leuprorelin Acetate 11.25 mg: Leuprorelin Acetate Injection Kit 11.25 mg, every 12 weeks subcutaneously, for up to at most 8 years. Participants received interventions as part of routine medical care.
  Interventions: Drug: Leuprorelin Acetate

INTERVENTIONS:
Drug: Leuprorelin Acetate — Leuprorelin Acetate Injection Kit
  Other Names: Leuplin SR for Injection Kit 11.25 mg

SUMMARY:
The purpose of this survey is to evaluate the long-term safety and efficacy of leuprorelin acetate injection kit 11.25 mg in patients with spinal and bulbar muscular atrophy (SBMA) in the routine clinical setting.

DETAILED DESCRIPTION:
The drug being tested in this survey is called leuprorelin acetate injection kit 11.25 mg. This injection kit is being tested to treat people who have SBMA.

This survey is an observational (non-interventional) study and will look at the long-term safety and efficacy of the leuprorelin acetate injection kit 11.25 mg in the routine clinical setting. The planned number of observed patients will be approximately 300.

This multi-center observational trial will be conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

* All SBMA patients who have been confirmed as receiving the drug

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SBMA patients treated with Leuprorelin Acetate Injection Kit 11.25 mg as part of routine medical care
Sampling Method: Probability Sample
Enrollment: 1890 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who had One or More Adverse Drug Reactions | Up to 1 Year
  Adverse drug reaction refers to adverse events related to administered drug. Percentage of participants who have the adverse drug reactions that occurred between initiation of treatment with the drug and 1 year after the start of treatment with the drug (or 3 months after the last dose of the drug if the treatment was discontinued within the first four doses) will be reported.
Percentage of Participants who had One or More Serious Adverse Events | Up to 1 Year
  Percentage of participants who have the serious adverse events that occurred between initiation of treatment with the drug and 1 year after the start of treatment with the drug (or 3 months after the last dose of the drug if the treatment was discontinued within the first four doses) will be reported.

SECONDARY OUTCOMES:
Percentage of Participants without Death Event | At final assessment point (up to 8 years)
  Percentage of participants without events of death at final assessment point (up to 8 years from initiation of treatment) will be reported.
Percentage of Participants without Pneumonia Requiring Hospitalization Event | At final assessment point (up to 8 years)
  Percentage of participants without events of pneumonia requiring hospitalization at final assessment point (up to 8 years from initiation of treatment) will be reported.
Percentage of Participants without Composite Events of Death and Pneumonia Requiring Hospitalization | At final assessment point (up to 8 years)
  Percentage of participants without composite events of death and pneumonia requiring hospitalization at final assessment point (up to 8 years from initiation of treatment) will be reported.
Percentage of Participants without Dysphagia Events | At final assessment point (up to 8 years)
  Percentage of participants without events of dysphagia at final assessment point (up to 8 years from initiation of treatment) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/5f6b60244db2bf003ab49792